CLINICAL TRIAL: NCT04194372
Title: Signature of the Risk Profile of Mortality in a Hospital Cohort of Patients With Metabolic Diseases
Acronym: INTEGRA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_08; 2019-A01727-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-04

CONDITIONS: Metabolic Disease
Keywords: Diabetic; CardioVascular Disease; morbi-mortality; Hospital Cohort
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, plasma, serum,nail appendage, hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metabolic Patient: Patients with a metabolic desease, defined as
  1. Metabolic Syndrom
  2. Diabetic
  3. Obese

SUMMARY:
Epidemiological studies are usually conducted in the general population in adults without complications or pathology at baseline. The results obtained are therefore often better designed for primary prevention use. The prediction of mortality risk in patients with complications and requiring hospital follow-up is less well known.

The study purpose is to determine a mortality risk profile in a hospital cohort of patients with pathologies associated with metabolic diseases.

Today the "multimaker" scores based on a panel of biomarkers - have significantly improved the discriminating power of prediction models existing in many pathologies. It is no longer a single biomarker that can improve risk prediction but a complete and cross-sectional profile that is sought after. We aim to establish a personalised mortality risk profile by combining clinical and biological parameters including metabolomics, genetics, transcriptomics and epigenomics by high throughput screening of biological samples.

DETAILED DESCRIPTION:
The prediction of the onset of diabetes and metabolic complications, especially cardiovascular, renal, or hepatic, is a major challenge to optimize the management of this disease.

Teams from the University Hospital of Lille have developed the Integra cohort study to identify the clinical and biological determinants of the occurrence of these complications and the mortality of patients with metabolic disorders.

The aim of the study is to identify clinico-biological determinants that are able to predict the occurence of death, cardiovascular events as well as hepatic or nephrotic one.

Follow-up data will be collected from National System of Health Data (SNDS) where data concerning hospitalisations, medical consultations and treatments are registered.

Biological samples are collected at baseline for a large OMICs analysis (metabolomics, genetics, transcriptomics and epigenomics) that would feed our predictive scoring system.

This project will allow us to describe new models of prediction of metabolic diseases and its complications, and to offer adapted and personalised methods of management, which can slow the progression of the disease and improve its prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic: antecedent - treatment - or glycemia> = 1.26 g / dl - or HbA1C> = 6.5% and or
* Obese: BMI> = 30 and or
* Metabolic syndrome defined AND
* Patient having given written consent to participate in the study or collection of the consent of the witness
* Social insured patient (excluding AME)
* Patient willing to comply with all procedures of the study and its duration AND

Patient also presenting a pathology among:

* Cardiology:

  * Coronary patient(history of myocardial infarction, coronary bypass, or coronary angioplasty or stenosis greater than 50% on an epicardial vessel documented on coronary angiography)
  * Patient with systolic or diastolic heart failure
  * Patient with atrial fibrillation
  * Patient with aortic stenosis (Vmax> 2.5 m / s)
  * Patient with high blood pressure
* neurology:

  * ischemic stroke
  * intracerebral hemorrhage
  * transient ischemic attack
* diabetology:

  * Obesity without diabetes
  * Diabetes T2
  * T1 diabetes
  * Monogenic Diabetes / MODY
  * African Diabetes
  * Diabetes secondary to pancreatopathy / liver cirrhosis
  * Diabetes post transplantation / post immunotherapy
  * Diabetes associated with Steinert's disease
* hepatology: hepatological pathology
* nephrology: nephrology

Exclusion Criteria:

* Unscheduled hospitalization less than 3 months old
* Ongoing treatment :

  * Cytotoxic chemotherapy
  * Radiotherapy
* HIV and / or HCV and / or active HBV infection
* OMS score> = 2
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pathologies associated with metabolic disease
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
number of death | at 10 years
  The number of patients dead according to national database

SECONDARY OUTCOMES:
Occurrence of macrovascular complications (composite criteria) | at 10 years
  composite criteria: cardiovascular death, myocardial infarction, stroke, coronary revascularization, peripheral revascularization, amputation)
hospitalization for heart failure | at 10 years
  The number of patients that has been hospitalized for heart failure since the end of the study according to national database
Occurence of renal microvasculare complications (composite criteria) | at 10 years
  composite criteria: renal transplantation, dialysis, GFR >60, Albuminuria
Occurrence of liver complications(composite endpoint) | at 10 years
  composite endpoint: hepatic fibrosis, cirrhosis, HCC, death from liver
Occurrence of hemorrhages measured by BARC >3 bleeding | at 10 years
  composite endpoint : CABG-related bleeding (Perioperative intracranial bleeding within 48 h / Reoperation after closure of sternotomy for the purpose of controlling bleeding / Transfusion of<5 U whole blood or packed red blood cells within a 48-hperiod / Chest tube output>=2L within a 24-h period)
  or Fatal Bleeding (Probable fatal bleeding; no autopsy or imaging confirmation butclinically suspicious / Definite fatal bleeding; overt bleeding or autopsy or imagingconfirmation)

CONTACTS AND LOCATIONS:
Overall Officials: François Pattou, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (3):
- France (3):
  - Ch Boulogne-Sur-Mer, Boulogne-sur-Mer
  - Hop Cardiologique Chr Lille, Lille
  - Hop Claude Huriez Chr Lille, Lille